CLINICAL TRIAL: NCT03471234
Title: LATIn American sTUdy to Investigate the Clinical Performance of Sirolimus-eluting Stent With Abluminal-only bioDEgradable Polymeric Coating (Inspiron TM) in the Treatment of Native Coronary Artery Lesions.
Brief Title: Latin America Real World Study With Inspiron Drug Eluting Stent - INSPIRON LATITUDE
Acronym: LATITUDE
Status: Completed | Type: Observational
Sponsor: Scitech Produtos Medicos Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: SCI-CO-01
Record Dates: First submitted 2018-03-05; First posted 2018-03-20 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; drug eluting stent; Inspiron
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Angioplasty — Inspiron Drug Eluting stent implantation

SUMMARY:
Prospective, multicenter, single arm registry to monitor post-market clinical outcomes of patients treated with Inspiron Sirolimus-Eluting Stent with Biodegradable Polymer.

DETAILED DESCRIPTION:
Prospective, multicenter, single arm registry to assess the safety and performance of Inspiron Sirolimus-Eluting Stent with Biodegradable Polymer for the treatment of "real world" patients.

ELIGIBILITY:
Inclusion Criteria:

* All individuals aged over 18 years who signed the informed consent and had lesions in native coronary arteries treated only with Inspiron Sirolimus-Eluting stent.

Exclusion Criteria:

* Saphenous vein grafts or Mammary lesions;
* Individuals who have been treated within the last 6 months with another stent;
* Acute myocardial infarction with ST segment elevation;
* Chronic Total Occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lesions in native coronary arteries measuring between 2.5 and 4.0 mm in diameter and 34 mm length treated only with Inspiron Sirolimus-Eluting Stent.
Sampling Method: Non-Probability Sample
Enrollment: 299 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
MACE (major cardiac events) | 12 months
  Major cardiac events (death, myocardial infarction, target vessel revascularization)

SECONDARY OUTCOMES:
Acute success | up to 24 hours
  Acute success measured by Angiography after stent implantation
Stent Thrombosis | 24 months
  Stent Thrombosis rate
MACE | 24 months
  Major cardiac events (death, myocardial infarction, target vessel revascularization)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coração - INCOR, São Paulo

IPD SHARING:
Plan to Share IPD: No